CLINICAL TRIAL: NCT01808222
Title: Transmolecular Imaging of Recurrent Prostate Carcinoma With Exploration of Genomic Markers Differences Between Local and Distant Recurrence
Brief Title: FACBC for Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David M. Schuster, MD (Other)
Responsible Party: Sponsor-Investigator, David M. Schuster, MD, MD, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00061518; FACBC2 (Other: Other)
Record Dates: First submitted 2013-03-05; First posted 2013-03-11 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- FACBC (Experimental): Participants receiving a bolus of anti-[18F]FACBC injected with PET-CT detection of cancer recurrence.
  Interventions: Drug: FACBC

INTERVENTIONS:
Drug: FACBC — Participants will receive a bolus of anti-[18F]FACBC injected IV over 1-2 minutes. The dosage will be approximately 10.0 millicuries (mCi) (3.70 x 108 becquerel (Bq)).
  Other Names: anti-[18F]FACBC

SUMMARY:
The investigators will perform a study with 25 patients in whom the investigators have a strong suspicion of prostate cancer that has returned to the body after having an initial treatment. The major goal of the investigation is to see whether anti-[18F] FACBC PET-CT and MRI imaging individually will be useful in the detection of local and extraprostatic recurrence of prostate cancer. Routine blood test will be done on the day of the FACBC scan and one week later as required by the FDA. All patients will undergo biopsy of the prostate as clinically appropriate per standard of care. If either the FACBC or MRI scans indicate cancer recurrence, the subject's cancer site(s) will also be biopsied as clinically appropriate.

DETAILED DESCRIPTION:
Prostate cancer is the most common solid tumor, with approximately 200,000 new cases diagnosed per year. Several different local therapies are available for treatment, including surgery and radiotherapy. Significant advances have been made which have improved the cancer control outcomes and treatment. Despite these significant advances, approximately 30% of patients treated with definitive local therapy experience recurrent disease. Recurrent (returning) disease usually displays rising Prostate-Specific Antigen (PSA) (a blood test for prostate cancer). The PSA level is often of limited use in differentiating local recurrence (i.e. recurrence in the prostate bed) from recurrence outside of the prostate bed (extra-prostatic recurrence). Imaging plays a central role in the detection of recurrent prostate carcinoma in the prostate bed and in the differentiation of prostatic from extraprostatic recurrence. There are newer methods of imaging such as magnetic resonance imaging (MRI) and positron emission tomography (PET) with molecular radiotracers that are currently under study for the imaging of post-therapy recurrence.

One PET radiotracer which has shown promise in the staging and restaging of patients with prostate carcinoma is anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid (anti-3-[18F]FACBC) which is a synthetic amino acid analog. FACBC demonstrated higher accuracy compared with other methods in the restaging of patients with suspected recurrent prostate carcinoma. FACBC has been tested in over 140 subjects in other studies in the Emory system including 128 subjects with prostate cancer.

The investigators will perform a study with 25 patients in whom the investigators have a strong suspicion of prostate cancer that has returned to the body after having an initial treatment. The major goal of the investigation is to see whether anti-[18F] FACBC PET-CT and MRI imaging individually will be useful in the detection of local and extraprostatic recurrence of prostate cancer. Routine blood test will be done on the day of the FACBC scan and one week later as required by the FDA.

All patients will undergo biopsy of the prostate as clinically appropriate per standard of care. If either the FACBC or MRI scans indicate cancer recurrence, the subject's cancer site(s) will also be biopsied as clinically appropriate. Biopsy of the suspected recurrence sites will be scheduled at the subjects' convenience as soon as possible after the scans.

Tissue obtained from the biopsy will undergo standard analysis to determine if prostate carcinoma cells are present. The secondary aim is to use left-over biopsy material to determine if there are genotypic differences between prostate carcinoma recurrence confined to the prostate bed and extraprostatic recurrence

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients will have been originally diagnosed with localized (Stage T1c, T2, or T3 ) prostate carcinoma and have undergone what was considered definitive non-prostatectomy therapy for localized disease.
3. In the case of cryotherapy, external beam radiation, or High-Intensity Focused Ultrasound (HiFU) the procedure will have occurred at least one year in the past. In the case of brachytherapy, treatment will have occurred at least 2 years in the past to eliminate patients with so-called "PSA bump."
4. Patient will have suspicion of recurrent prostate carcinoma as defined by: the Radiation Therapy Oncology Group (RTOG) - American Society for Therapeutic Radiology and Oncology (ASTRO) Phoenix criteria of nadir PSA +2, and absolute PSA ≥ 4.0 ng/ml.with any doubling time (DT) or with PSA 2.0-3.99 ng/ml with DT ≤10 months
5. Ability to lie still for PET scanning
6. Patients must be able to provide written informed consent.

Exclusion Criteria:

1. Age less than 18.
2. Greater than T3 disease in past and/or treated with prostatectomy.
3. Less than 1 year since cryotherapy,external beam radiation therapy, or HiFU or 2 years since brachytherapy..
4. Does not meet above criteria of suspicious PSA elevation
5. Inability to lie still for PET scanning
6. Cannot provide written informed consent.
7. Bone scan findings characteristic for metastatic prostate carcinoma
8. Less than 1 month since any prior prostate biopsy (to decrease false positive uptake from inflammation).

   -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Akin-Akintayo O, Tade F, Mittal P, Moreno C, Nieh PT, Rossi P, Patil D, Halkar R, Fei B, Master V, Jani AB, Kitajima H, Osunkoya AO, Ormenisan-Gherasim C, Goodman MM, Schuster DM. Prospective evaluation of fluciclovine (18F) PET-CT and MRI in detection of recurrent prostate cancer in non-prostatectomy patients. Eur J Radiol. 2018 May;102:1-8. doi: 10.1016/j.ejrad.2018.02.006. Epub 2018 Feb 24. PMID 29685521

RESULTS

PARTICIPANT FLOW:
Groups:
- FACBC: Participants receiving a bolus of anti-[18F]FACBC injected with positron emission tomography (PET)-computerized tomography (CT) (PET-CT) and a multiparametric MRI (mpMR) for detection of cancer recurrence.
Period: Overall Study
Arm/Group | FACBC
Started | 25
Completed Fluciclovine PET-CT Scan | 25
Completed mpMR Scan | 24
Completed | 24
Not Completed | 1
Not completed — mpMR scan was not performed | 1

BASELINE CHARACTERISTICS:
Population: Participants completing both scans are included in the baseline analysis.
Groups:
- FACBC: Participants receiving a bolus of anti-[18F]FACBC injected with PET-CT and a multiparametric MRI for detection of cancer recurrence.
Arm/Group | FACBC
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24
PET-MR Interval [Median (Full Range); unit: days] | 7.5 [0 to 29]
Prior prostate cancer therapy [Count of Participants; unit: Participants]
  Brachytherapy alone | 3
  Brachytherapy with one | 8
  Brachytherapy as part of 3+ treatments | 5
  Radiotherapy alone | 3
  3+ Other Treatment Modalities | 2
  Proton Therapy | 1
  Cryotherapy alone | 1
  Cryotherapy plus hormonal therapy | 1
Prostate-Specific Antigen (PSA) [Mean (Standard Deviation); unit: Nanograms per milliliter (ng/ml)] | 8.5 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: The Presence of Cancer Tissue Inside of the Prostate Bed
Description: Participants had a fluciclovine PET-CT scan and a multiparametric magnetic imaging (mpMR) scan. The scans were read by experts (two for the PET-CT scans and two more for the mpMR scans) and the accuracy of each imaging technique was assessed by comparing the interpretations of the imaging to biopsy results. The degree of confidence of interpretation of each reader was recorded on a 5-point Likert scale where:
  1. = definitely benign
  2. = probably benign
  3. = equivocal
  4. = probably malignant
  5. = definitely malignant For this analysis, scores of 4 or 5 were considered positive and scores of 1-3 were considered negative for malignant prostate disease.
Time Frame: Up to 43 months
Population: The population assessed in this analysis includes participants with sufficient proof for the absence of presences of prostate disease (22 out of 24 participants who received both scans). The remaining two had no biopsy or had insufficient follow-up information to reach a consensus about disease status.
Measure: Count of Participants; unit: Participants
Arm/Group | FACBC
Number analyzed (Participants) | 22
Participants
  PET-CT Readers 1 and 2: True Positivies | 13
  PET-CT Readers 1 and 2: False Positives | 8
  PET-CT Readers 1 and 2: True Negatives | 1
  PET-CT Readers 1 and 2: False Negatives | 0
  mpMR Reader 1: True Positivies | 5
  mpMR Reader 1: False Positives | 4
  mpMR Reader 1: True Negatives | 5
  mpMR Reader 1: False Negatives | 8
  mpMR Reader 2: True Positivies | 2
  mpMR Reader 2: False Positives | 2
  mpMR Reader 2: True Negatives | 7
  mpMR Reader 2: False Negatives | 11

2. Primary Outcome: The Presence of Cancer Tissue Outside of the Prostate Bed
Description: as for outcome 1
Time Frame: Up to 43 months
Population: The population assessed in this analysis includes participants with sufficient proof for the absence of presences of prostate disease (18 out of 24 participants who received both scans).
Measure: Count of Participants; unit: Participants
Arm/Group | FACBC
Number analyzed (Participants) | 18
Participants
  PET-CT Readers 1 and 2: True Positives | 7
  PET-CT Readers 1 and 2: False Positives | 1
  PET-CT Readers 1 and 2: True Negatives | 9
  PET-CT Readers 1 and 2: False Negatives | 1
  mpMR Reader 1: True Positives | 4
  mpMR Reader 1: False Positives | 3
  mpMR Reader 1: True Negatives | 7
  mpMR Reader 1: False Negatives | 4
  mpMR Reader 2: True Positives | 6
  mpMR Reader 2: False Positives | 2
  mpMR Reader 2: True Negatives | 8
  mpMR Reader 2: False Negatives | 2

ADVERSE EVENTS:
Time Frame: Adverse events related to the study procedures were collected from the time a participant consented to take part in the trial through all study related procedures (up to 29 days, which is the maximum number of days between a participant receiving both imaging tests). Adverse events related to the study procedures were not expected.
Arm/Group | FACBC
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT01808222/Prot_SAP_000.pdf